CLINICAL TRIAL: NCT02285998
Title: Comparison of the Protective Efficacy of Flublok® Quadrivalent Versus Licensed Inactivated Influenza Vaccine (IIV4) in Healthy, Medically Stable Adults ≥50 Years of Age
Brief Title: Protective Efficacy of Flublok® Quadrivalent Versus Licensed Inactivated Influenza Vaccine in Adults ≥50 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Protein Sciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PSC12
Record Dates: First submitted 2014-10-27; First posted 2014-11-07 (Estimated); Results first posted 2016-10-04 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-09

CONDITIONS: Influenza
Keywords: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flublok Quadrivalent Influenza Vaccine (Experimental): Intramuscular injection of vaccine containing 4 x 45µg (180µg total) of each recombinant hemagglutinin (rHA) derived from influenza A/H1N1 and A/H3N2 and two lineages of influenza B viruses identified for the season in which the trial is conducted in a total volume of 0.5 mL
  Interventions: Biological: Flublok Quadrivalent Influenza Vaccine
- Inactivated Influenza Vaccine (Active Comparator): Intramuscular injection of vaccine contains 4 x 15µg (60µg total) of HA derived from the same influenza A/H1N1 and A/H3N2 and influenza B strains in a total volume of 0.5mL.
  Interventions: Biological: Inactivated Influenza Vaccine

INTERVENTIONS:
Biological: Flublok Quadrivalent Influenza Vaccine — Intramuscular injection of vaccine
  Arms: Flublok Quadrivalent Influenza Vaccine
Biological: Inactivated Influenza Vaccine — Intramuscular injection of vaccine
  Arms: Inactivated Influenza Vaccine

SUMMARY:
The goal of this study is to establish that Flublok Quadrivalent is non-inferior to fully licensed (traditional approval status) quadrivalent inactivated influenza vaccine (IIV4) in protecting against laboratory-confirmed clinical influenza disease in the ≥50 year age population.

DETAILED DESCRIPTION:
The goal of this study is to establish that Flublok Quadrivalent is non-inferior to fully licensed (traditional approval status) quadrivalent inactivated influenza vaccine (IIV4) in protecting against laboratory-confirmed clinical influenza disease in the ≥50 year age population. Real-time Polymerase Chain Reaction (rtPCR) will be used to confirm influenza infection and to type the strains involved, as molecular methodologies have been demonstrated to be more sensitive than other more traditional methodologies, e.g. culture. For rtPCR-positive clinical samples, reserved aliquots will be processed for culture, so that antigenic similarity to the HA present in study vaccines can be tested.

In various clinical studies the investigators demonstrated that the immune response against the influenza A viruses is improved as a result of the higher hemagglutinin content. Furthermore, influenza virus disease and hospitalization associated with influenza-related illness in older adults (> 50 years) was considerably reduced (90%) following vaccination with TIV, even though the circulating influenza A strain was antigenically dissimilar to that in the vaccine. However, more recently Skowronski et al. reported that the low influenza vaccine effectiveness in 2012-2013 was not associated with antigenic drift but was instead related to mutations in the egg-adapted H3N2 vaccine strain. Flublok manufactured using recombinant technology does not contain the mutations responsible for the reported lower effectiveness and may thus offer improved protection when mutations such as those described are induced in the process of adapting the influenza virus to growth in eggs.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory adults aged 50 and older.
2. Medically stable, as determined by medical history and targeted physical examination. "Medically stable" is defined as no change in diagnoses or chronic medications (dose or class) for medical reasons in the 3 months prior to study.
3. Absence of underlying conditions that make participation in the study contrary to the subject's best interest.
4. Able to understand and comply with planned study procedures.
5. Provides written informed consent prior to initiation of any study procedure.

Exclusion Criteria:

1. Known contraindication to either study vaccine (see product package inserts)
2. Receipt of any other influenza vaccine within 180 days prior to enrollment in this study.
3. Underlying disease or ongoing therapy that might cause immunocompromise, e.g. cytotoxic agents or supraphysiologic doses of corticosteroids, such that response to vaccination might be sub-optimal.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9003 (Actual)
Dates: Start 2014-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (38):
- United States (38):
  - Coastal Clinical Research, Mobile, Alabama
  - Clinical Research Consortium Arizona, Tempe, Arizona
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - Northern California Clinical Research Center, Redding, California
  - Benchmark Research - Sacramento, Sacramento, California
  - Benchmark Research - San Francisco, San Francisco, California
  - Lynn Institute of the Rockies, Colorado Springs, Colorado
  - Clinical Research Consulting, Milford, Connecticut
  - Clinical Research of South Florida, Coral Gables, Florida
  - Avail Clinical Research, DeLand, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Meridian Research, Savannah, Georgia
  - ACR - Boise, Meridian, Idaho
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Central Kentucky Research Associates, Lexington, Kentucky
  - Benchmarch Research - New Orleans, Metairie, Louisiana
  - ActivMed Practices & Research, Methuen, Massachusetts
  - Center for Pharmaceutical Research, Kansas City, Missouri
  - Meridian Research, Bellevue, Nebraska
  - Meridian Research, Norfolk, Nebraska
  - Meridian Clinical Research, Omaha, Nebraska
  - Clinical Research Consortium-Nevada, Las Vegas, Nevada
  - ActivMed Practices & Research, Newington, New Hampshire
  - Regional Clinical Research, Inc., Endwell, New York
  - Rochester Clinical Research, Rochester, New York
  - Wake Research, Raleigh, North Carolina
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Lynn Institute of Norman, Norman, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Meridian Research, Dakota Dunes, South Dakota
  - Clinical Research Associates, Nashville, Tennessee
  - Benchmark Reseach, Austin, Texas
  - Benchmark Research - Fort Worth, Fort Worth, Texas
  - Benchmark Research - San Angelo, San Angelo, Texas
  - Jean Brown Research, Salt Lake City, Utah
  - Clinical Research Associates of Tidewater, Norfolk, Virginia

REFERENCES:
- [Derived] Dunkle LM, Izikson R, Patriarca P, Goldenthal KL, Muse D, Callahan J, Cox MMJ; PSC12 Study Team. Efficacy of Recombinant Influenza Vaccine in Adults 50 Years of Age or Older. N Engl J Med. 2017 Jun 22;376(25):2427-2436. doi: 10.1056/NEJMoa1608862. PMID 28636855

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Excludes 40 subjects who received randomization numbers, but who either withdrew prior to vaccination (n=15) or for whom the vaccine received could not be verified (n=25; 12 assigned to Flublok quadrivalent and 13 assigned to IIV4).
Period: Overall Study
Arm/Group | Flublok Quadrivalent Influenza Vaccine | Inactivated Influenza Vaccine
Started | 4474 | 4489
Completed | 4228 | 4236
Not Completed | 246 | 253
Not completed — Adverse Event | 9 | 8
Not completed — Physician Decision | 1 | 2
Not completed — Lost to Follow-up | 176 | 172
Not completed — Withdrawal by Subject | 53 | 61
Not completed — Other Reasons | 7 | 10

BASELINE CHARACTERISTICS:
Population: The safety population included all randomized subjects who received known study vaccine and for whom some safety data were available after administration of vaccine.
Groups:
- Total: Total of all reporting groups
Arm/Group | Flublok Quadrivalent Influenza Vaccine | Inactivated Influenza Vaccine | Total
Number analyzed (Participants) | 4328 | 4344 | 8672
Age, Customized [Number; unit: participants]
  50-64 years | 2569 | 2617 | 5186
  65-74 years | 1234 | 1254 | 2488
  75 years and older | 525 | 473 | 998
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2532 | 2537 | 5069
  Male | 1796 | 1807 | 3603

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With rtPCR-confirmed Influenza-Like Illness
Description: rtPCR-confirmed, protocol-defined Influenza-Like Illness (ILI) caused by any influenza strain that begins at least 14 days post-vaccination
Time Frame: 14 days post vaccination through and up to 32 weeks post vaccination
Population: The efficacy population includes all randomized subjects who received study vaccine and provided any follow-up for ILI beginning at least 14 days following vaccine administration.
Measure: Number; unit: participants
Arm/Group | Flublok Quadrivalent Influenza Vaccine | Inactivated Influenza Vaccine
Number analyzed (Participants) | 4303 | 4301
participants | 96 | 138
Statistical Analysis 1: Comparison: Flublok Quadrivalent Influenza Vaccine vs Inactivated Influenza Vaccine; The primary efficacy analysis was based on the numbers of protocol-defined influenza-like illnesses with rtPCR-positive nasopharyngeal swabs detecting influenza virus of any strain. The Relative Vaccine Efficacy was 30% (10, 47). Non-inferiority would be concluded if the lower bound of the 95% CI for rVE was > -20%. Superiority of RIV4 in a pre-specified exploratory analysis required that the lower bound of the two-sided 95% CI of rVE be > +9%; Test type: Non-Inferiority or Equivalence — The sample size required to achieve 80% power was calculated based on a one-sided alpha level of 0.025 and an attack rate of 2% in the IIV4 and 1.53% for the Flublok groups respectively; Relative Vaccine Efficacy (rVE) = 30, 95% CI 2-sided [10 to 47]

2. Secondary Outcome: Number of Participants With Culture-confirmed Influenza-Like Illness
Description: Culture-confirmed protocol-defined Influenza-Like Illness (ILI) that begins at least 14 days post-vaccination caused by an influenza strain (identified from the same clinical sample) antigenically matched to those strains represented in the study vaccines.
  Protocol-defined ILI is defined as at least one of the following respiratory symptoms accompanied by at least one of the following systemic symptoms:
  Respiratory symptoms: sore throat, cough, sputm production, wheezing, difficulty breathing Systemic symptoms: fever, chills (shivering), tiredness (fatigue), headache, myalgia (muscle ache)
Time Frame: 14 days post vaccination through and up to 32 weeks post vaccination
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Flublok Quadrivalent Influenza Vaccine | Inactivated Influenza Vaccine
Number analyzed (Participants) | 4303 | 4301
participants | 58 | 101

3. Secondary Outcome: Number of Participants With Culture-confirmed CDC-defined Influenza-Like Illness
Description: Culture-confirmed CDC-defined Influenza-Like Illness (ILI) that begins at least 14 days post-vaccination caused by an influenza strain (identified from the same clinical sample) antigenically matched to those in the study vaccines.
  CDC-defined ILI is defined as body temperature ≥100°F accompanied by cough and/or sore throat.
Time Frame: 14 days post vaccination through and up to 32 weeks post vaccination
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Flublok Quadrivalent Influenza Vaccine | Inactivated Influenza Vaccine
Number analyzed (Participants) | 4303 | 4301
participants | 38 | 64

4. Secondary Outcome: Number of Participants With rtPCR-confirmed CDC-defined Influenza-Like Illness
Description: rtPCR-confirmed CDC-defined ILI that begins at least 14 days post-vaccination caused by any influenza strain.
Time Frame: 14 days post vaccination through and up to 32 weeks post vaccination
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Flublok Quadrivalent Influenza Vaccine | Inactivated Influenza Vaccine
Number analyzed (Participants) | 4303 | 4301
participants | 54 | 83

5. Secondary Outcome: Percentage of Participants With Seroconversion
Description: Seroconversion rates (SCR) for all four antigens in a preselected subset of subjects.
Time Frame: Days 0 through 28
Population: The immunogenicity population includes all randomized subjects at the specific study sites pre-selected for serology who received study vaccine and provided serum samples on Days 0 and 28 for serologic testing.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Flublok Quadrivalent Influenza Vaccine | Inactivated Influenza Vaccine
Number analyzed (Participants) | 314 | 300
percentage of participants
  A/California | 44.9 [39.3 to 50.6] | 49.0 [43.2 to 54.8]
  A/Texas | 54.5 [48.8 to 60.1] | 43.3 [37.6 to 49.1]
  B/Massachusetts | 38.9 [33.4 to 44.5] | 38.3 [32.8 to 44.1]
  B/Brisbane | 21.0 [16.6 to 25.9] | 34.3 [29.0 to 40.0]

6. Secondary Outcome: Number of Participants With Local Injection Site Reactogenicity
Description: Solicited events of injection site reactogenicity reported during Day 0-7.
Time Frame: Days 0 through 7
Population: Solicited local reactogenicity events include subjects who recorded any injection site reaction data.
Measure: Number; unit: participants
Arm/Group | Flublok Quadrivalent Influenza Vaccine | Inactivated Influenza Vaccine
Number analyzed (Participants) | 4307 | 4319
participants | 1621 | 1745

7. Secondary Outcome: Number of Participants With Unsolicited Adverse Events
Description: Unsolicited adverse events reported in the 28 days following vaccine administration.
Time Frame: Days 0 through 28
Population: The safety population includes all randomized and vaccinated subjects who provided any safety data (solicited or unsolicited) following administration of study vaccine.
Measure: Number; unit: participants
Arm/Group | Flublok Quadrivalent Influenza Vaccine | Inactivated Influenza Vaccine
Number analyzed (Participants) | 4328 | 4344
participants | 1345 | 1355

8. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Medically-attended Adverse Events (MAEs)
Description: Serious adverse events (SAEs) and medically-attended adverse events (MAEs) occurring during the period of follow-up through the influenza season (at least 6 months post-vaccination).
  A MAE is an event that prompts an unplanned visit to a medical professional for diagnosis and/or treatment.
Time Frame: Day 0 through and up to 32 weeks post vaccination
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Flublok Quadrivalent Influenza Vaccine | Inactivated Influenza Vaccine
Number analyzed (Participants) | 4328 | 4344
participants
  SAEs | 145 | 132
  MAEs | 774 | 785

9. Secondary Outcome: Measure of Post-vaccination HAI GMTs
Description: GMT titers for all four antigens in a preselected subset of subjects.
Time Frame: Days 0 through 28
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Flublok Quadrivalent Influenza Vaccine | Inactivated Influenza Vaccine
Number analyzed (Participants) | 314 | 300
titer
  Day 0 - A/California | 45 [38 to 52] | 49 [42 to 57]
  Day 28 - A/California | 194 [167 to 226] | 224 [197 to 255]
  Day 0 - A/Texas | 88 [74 to 104] | 100 [84 to 119]
  Day 28 - A/Texas | 530 [470 to 597] | 366 [325 to 412]
  Day 0 - B/Massachusetts | 17 [15 to 20] | 18 [16 to 21]
  Day 28 - B/Massachusetts | 56 [49 to 64] | 58 [51 to 66]
  Day 0 - B/Brisbane | 14 [12 to 15] | 15 [13 to 16]
  Day 28 - B/Brisbane | 30 [26 to 34] | 44 [39 to 50]

10. Secondary Outcome: Number of Participants With Systemic Reactogenicity
Description: Solicited events of systemic reactogenicity reported during Day 0-7.
Time Frame: Days 0 through 7
Population: Solicited systemic reactogenicity events include subjects who recorded any systemic reaction data.
Measure: Number; unit: participants
Arm/Group | Flublok Quadrivalent Influenza Vaccine | Inactivated Influenza Vaccine
Number analyzed (Participants) | 4306 | 4318
participants | 1077 | 1106

ADVERSE EVENTS:
Time Frame: From time vaccination until the end of the influenza season (~6 months).
Arm/Group | Flublok Quadrivalent Influenza Vaccine | Inactivated Influenza Vaccine
Serious Adverse Events (participants affected / at risk) | 145/4328 | 132/4344
Other Adverse Events (participants affected / at risk) | 1122/4328 | 1206/4344
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Flublok Quadrivalent Influenza Vaccine (N=4328) | Inactivated Influenza Vaccine (N=4344)
Pneumonia (Infections and infestations) | 6 | 6
Bronchitis (Infections and infestations) | 2 | 3
Diverticulitis (Infections and infestations) | 2 | 2
Influenza (Infections and infestations) | 1 | 3
Urinary tract infection (Infections and infestations) | 2 | 2
Cellulitis (Infections and infestations) | 0 | 3
Appendicitis (Infections and infestations) | 1 | 1
Lung Infection (Infections and infestations) | 1 | 1
Osteomyelitis (Infections and infestations) | 1 | 1
Pyelonephritis (Infections and infestations) | 1 | 1
Abscess intestinal (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Endocarditis staphylococcal (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1
Eye abscess (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 0 | 1
Osteomyelitis acute (Infections and infestations) | 0 | 1
Osteomyelitis chronic (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0
Salmonellosis (Infections and infestations) | 1 | 0
Urinary tract infection fungal (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 6 | 3
Myocardial infarction (Cardiac disorders) | 4 | 3
Angina pectoris (Cardiac disorders) | 2 | 2
Cardiac failure congestive (Cardiac disorders) | 2 | 2
Angina unstable (Cardiac disorders) | 2 | 1
Coronary artery disease (Cardiac disorders) | 2 | 1
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 0 | 1
Coronary artery insufficiency (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Coronary artery thrombosis (Cardiac disorders) | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 8 | 7
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 5 | 6
Transient ischaemic attack (Nervous system disorders) | 3 | 2
Syncope (Nervous system disorders) | 1 | 3
Convulsion (Nervous system disorders) | 1 | 1
Embolic stroke (Nervous system disorders) | 2 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Lacunar infarction (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 1
Myelomalacia (Nervous system disorders) | 1 | 0
Sinus headache (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Thalamic infarction (Nervous system disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Cyclic vomiting syndrome (Gastrointestinal disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Volvulus (Gastrointestinal disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Abdominal wall neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rhabdomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chest pain (General disorders) | 7 | 6
Death (General disorders) | 2 | 1
Non-cardiac chest pain (General disorders) | 3 | 0
Asthenia (General disorders) | 0 | 1
Drug withdrawal syndrome (General disorders) | 0 | 1
Hernia obstructive (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 2
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Stab wound (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0
Aortic aneurysm rupture (Vascular disorders) | 0 | 1
Aortic dissection (Vascular disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 2 | 0
Abdominal hernia repair (Surgical and medical procedures) | 1 | 0
Alcohol detoxification (Surgical and medical procedures) | 0 | 1
Drug detoxification (Surgical and medical procedures) | 0 | 1
Gastric bypass (Surgical and medical procedures) | 1 | 0
Hernia repair (Surgical and medical procedures) | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 0 | 1
Inguinal hernia repair (Surgical and medical procedures) | 0 | 1
Intestinal resection (Surgical and medical procedures) | 1 | 0
Joint surgery (Surgical and medical procedures) | 1 | 0
Rotator cuff repair (Surgical and medical procedures) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 3 | 1
Urinary retention (Renal and urinary disorders) | 2 | 0
Bladder outlet obstruction (Renal and urinary disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Renal necrosis (Renal and urinary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Hepatic haemorrhage (Hepatobiliary disorders) | 0 | 1
Hepatitis alcoholic (Hepatobiliary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Uterine disorder (Reproductive system and breast disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0
Haematocrit decreased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 1 | 0
Troponin increased (Investigations) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Flublok Quadrivalent Influenza Vaccine (N=4328) | Inactivated Influenza Vaccine (N=4344)
Cough (Respiratory, thoracic and mediastinal disorders) | 226 | 253
Influenza like illness (General disorders) | 186 | 199
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 178 | 177
Headache (Nervous system disorders) | 143 | 145
Upper respiratory tract infection (Infections and infestations) | 129 | 156
Fatigue (General disorders) | 106 | 100
Myalgia (Musculoskeletal and connective tissue disorders) | 95 | 79
Productive cough (Respiratory, thoracic and mediastinal disorders) | 59 | 97

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No